CLINICAL TRIAL: NCT04300153
Title: The Effect of Erector Spinae Plane Block on Quality of Recovery and Postoperative Analgesia of Patients Undergoing Inguinal Hernia Repair: Randomized, Controlled, Double Blinded Trial
Brief Title: The Effect of Erector Spinae Plane Block on Quality of Recovery and Postoperative Analgesia After Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Başak Altıparmak (Other)
Collaborators: Muğla Sıtkı Koçman University (Other)
Responsible Party: Sponsor-Investigator, Başak Altıparmak, Assoc Prof, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-II
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Pain; Inguinal Hernia; Acute Pain
Keywords: erector spinae plane block; inguinal hernia; interfascial plane; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP Group (Experimental): At the end of the skin closure, patients will be positioned in lateral decubitis and unilateral ESP block will be performed with single injection of 30 ml 0.25% bupivacaine at the level of T12 transverse process. All patients will receive intravenous (iv) paracetamol 1000 mg at the arrival to the recovery room. The dosage will be repeated at every 8-hours interval.
  Interventions: Procedure: ESP Block; Other: Global Quality of Recovery-15 score; Other: Standard Pain Followup and Monitorization
- Control Group (Sham Comparator): At the end of the skin closure, patients will be positioned in lateral decubitis and unilateral ESP block will be performed with single injection of 30 ml normal saline at the level of T12 transverse process. All patients will receive intravenous (iv) paracetamol 1000 mg at the arrival to the recovery room. The dosage will be repeated at every 8-hours interval.
  Interventions: Procedure: ESP Block; Other: Global Quality of Recovery-15 score; Other: Standard Pain Followup and Monitorization

INTERVENTIONS:
Procedure: ESP Block — At the end of the skin closure, patients will be positioned in lateral decubitis with the involved site lying superiorly. A convex ultrasound probe will be placed over the transverse process of T12 vertebra in longitudinal axis and an 80- mm 21-gauge needle will be inserted in the plane view under aseptic conditions. A unilateral ESP block will be performed with 30 ml 0.25% bupivacaine into the interfascial plane between erector spinae muscle and T12 transverse process
Other: Global Quality of Recovery-15 score — Global Quality of Recovery-15 score (QoR-15) will be recorded prior to the surgery and at the postoperative 24th hour.
Other: Standard Pain Followup and Monitorization — Numeric Rating Scale score will be recorded at the 1.-2.-4.-6.-8.-12.-24.hours. If Numerical Rating Scale score will be equal to or over 4, iv dexketoprofen 50 mg will be applied as rescue analgesic. Numerical Rating Scale scores, the rescue analgesic need and the time for first mobilization of the patient will be recorded and kept in a statistical evaluation.

SUMMARY:
Inguinal hernia repair (IHR) is one of the most commonly performed operations in general surgery practice. Different pharmacological approaches and interfascial plane blocks are used to control postoperative pain. Erector spinae plane (ESP) block is a relatively new interfascial plane block which was reported to be effective in different types of surgeries. In this study, the primary aim is to assess the effect of ESP on recovery of patients following open IHR surgery.

DETAILED DESCRIPTION:
Inguinal hernia repair (IHR) is one of the most commonly performed operations in general surgery practice. Unfortunately, 40% of the patients experience moderate-to-severe acute pain in the early period. Erector spinae plane (ESP) block is a relatively new interfascial plane block which was described in 2016. In this prospective, controlled trial, the primary hypothesis is that ultrasound-guided unilateral ESP block will provide an increase in the quality of recovery-15 scores which will be assessed at the postoperative 24th hour following open IHR surgery. The secondary hypothesis is that ESP block will reduce postoperative pain scores, need for rescue analgesia and time to first mobilization.The study will be conducted as a single-center, prospective, randomized, controlled, double-blinded trial in a university hospital. Patients scheduled for an elective unilateral open IHR under spinal anesthesia, will be screened for enrollment to the study. At the end of the operation, patients will be randomized to receive a unilateral ESP block with 30 ml of 0.25% bupivacaine or 30 ml of normal saline at the level of T12 vertebrae. A blinded anesthesiologist will collect outcome measures in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I-II
* Elective unilateral open inguinal hernia repair under spinal anesthesia

Exclusion Criteria:

* Coagulation disorder
* Known allergy to study drugs
* Chronic opioid use
* Infection at the injection site
* Use of pain medications
* Psychologic disorder or inability to cooperate Quality of Recovery-15 (QoR-15) test
* Preoperative pain related to inguinal hernia NRS > 4/10

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-08 (Actual)

PRIMARY OUTCOMES:
Global Quality of Recovery-15 score | Postoperative 24th hour
  Global quality of recovery (QoR) score which will be measured by using 15-item QoR-15 questionnaire. This questionnaire covers a total of 15 questions under five clinical dimensions of health; physical comfort (five-item), emotional status (four-item), psychological support (two-item), physical independence (two-item) and pain (two-item)

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) | 24 hours
  A blinded anesthesiologist will assess postoperative pain of the patients during resting and movement at the 1st, 2nd, 4th, 6th, 8th, 12th and 24th hours by using 11-point Numerical Rating Scale which ranges from '0' (means no pain) to '10' (means worst pain imaginable).
Rescue analgesia | 24 hours
  If Numerical Rating Scale score of the patient is equal to or over 4, iv dexketoprofen 50 mg will be applied as rescue analgesic. Total rescue analgesia need will be recorded.
Mobilization time | 24 hours
  If the patient walks with or without help, it will be accepted as the first mobilization. The motor block duration and time for the first mobilization of the patient will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Başak Altıparmak, Principal Investigator — Muğla Sıtkı Koçman University Medical Faculty
Locations (1):
- Muğla Sıtkı Koçman University, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
via email